CLINICAL TRIAL: NCT01897623
Title: Prevalence and Screening of Abdominal Aortic Aneurysms Among Men With Coronary Artery Disease
Acronym: CAD-AAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Collaborators: Kuopio University Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Ville Vänni, General surgeon, North Karelia Central Hospital
Purpose: Screening
Other Study IDs: AAA-CAD-02
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound of aorta (Other)
  Interventions: Other: ultrasound of aorta

INTERVENTIONS:
Other: ultrasound of aorta

SUMMARY:
The purpose of this study is to investigate the prevalence of abdominal aortic aneurysms (AAA) among male patients with coronary artery disease (CAD) verified in coronary angiography. Ethiology of AAA is known to be common with atherosclerotic arterial diseases (coronary artery disease, peripheral artery disease and carotid artery disease), so the hypothesis is that AAA should be more common among these CAD patients, thus making screening of these patients (for AAA) more cost-efficient.

Study will be carried out as a multi-center prospective screening study. Data will be collected in North Karelia Central Hospital, Kuopio University Hospital and Tampere University Hospital. Data consists of 200 consecutive coronary angiography patients in each hospital, resulting in 600 patients in total. All male patients with diagnosed CAD will be recruited for the study and screened for AAA with ultrasound. Nevertheless, patients with previously known AAA will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with coronary artery disease

Exclusion Criteria:

* Patient's denial to participate
* Female Gender
* Already diagnosed or treated abdominal aortic aneurysm

Sex: Male
Age Groups: Child, Adult, Older Adult
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum diameter (mm) of abdominal aorta (outer-to-outer wall) in ultrasound | upon screening

CONTACTS AND LOCATIONS:
Locations (1):
- North Carelia Central Hospital, Joensuu, Pohjois-Karjala, Finland